CLINICAL TRIAL: NCT02425436
Title: Effects of Oral Ginkgo Biloba Extract on Pregnancy Complicated by Asymmetrically Intrauterine Growth Restriction: a Double-blinded Randomized Placebo-controlled Trial
Brief Title: Role of Ginkgo Biloba Extract in IUGR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamad sayed abdellah, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tibonina/ IUGR
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Intrauterine Growth Restriction (IUGR)
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginkgo Biloba Extract group (Active Comparator): This group received Ginko Biloba, two tablets per day
  Interventions: Drug: Ginkgo Biloba Extract
- Placebo group (Placebo Comparator): This group received placebo two tablets per day .
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ginkgo Biloba Extract
  Arms: Ginkgo Biloba Extract group
Other: Placebo
  Arms: Placebo group

SUMMARY:
The use of herbal medicinal products is increasing enormously in recent years, mainly among women, who use them for the most varied purposes, such as in menstrual problems, menopausal symptoms, mood disturbances and to strengthen their bones. Most of these benefits are due to the flavonoids present in these products. These flavonoids have anticarcinogenic, antiviral, antioxidant and antiinflammatory activities, as well as being used in the treatment of osteoporosis, menopausal symptoms and cardiovascular diseases . Besides the benefits from the consumption of flavonoids, little is known about their safety and potentially harmful toxic effects, such as mutagenicity and genotoxicity which might occur if taken in large doses . Safety of Ginkgo biloba during pregnancy or lactation was not criticized in literature. Roasted and raw ginkgo seed were not reported in the evidence-based medicine literature as being either safe or contraindicated in pregnancy or lactation. A higher incidence of postpartum hemorrhage was reported in the literature when associated with a 3-month ingestion of Ginkgo Biloba extract. Flavonoids are components of Ginkgo biloba L. (Ginkgoaceae), a medicinal plant widely used by the population . G. biloba has its origin in China, Korea and Japan where its fruits and leaves have been used as food and medicine for a long time.

The extract of G. biloba (EGb) is composed of different terpene trilactones, i.e., ginkgolides A, B, C, J and bilobalide, many flavonol glycosides, biflavones and alkylphenols . The major flavonoids in the extract are kaempferol, quercetin and isorhamnetin] whose metabolites were found in the blood of rats and in human urine after oral administration of EGb. Due to its actions as an anti-inflammatory and antioxidant, EGb has been largely used in the treatment of Alzheimer's disease, pre-menstrual syndrome, cerebrovascular insufficiency and peripheral arterial occlusive disease . In folk medicine, EGb is used as a vermifuge, to induce labor, for the treatment of bronchitis, chronic rhinitis, chilblains, arthritis and edema . The aim of this study was to evaluate the effect of oral supplementation of Ginkgo Biloba extract on the fetal weight as well as feto-maternal blood flow in cases of intrauterine growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their third trimester (28-30 weeks of gestation).
* Pregnant women whose pregnancy was complicated with intra uterine growth restriction (IUGR).
* Normal Doppler indices in uterine, umbilical and middle cerebral arteries at time of recruitment.

Exclusion Criteria:

* Multiple pregnancies,
* Hypertension,
* Fetal congenital anomalies,
* Previous history of congenital anomalies or chromosomal abnormalities.
* Diabetes Mellitus
* Premature pre-labor rupture of membranes
* Antepartum hemorrhage

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Fetal weight (gm) | one and half year

SECONDARY OUTCOMES:
Doppler blood flow changes in uterine arteries indices | one and half year
Doppler blood flow changes in umbilical arteries indices | one and half year
Doppler blood flow changes in middle cerebral artery indices | one and half year

IPD SHARING:
Plan to Share IPD: Yes